CLINICAL TRIAL: NCT03267290
Title: A Prospective Clinical Study for Comparing Diagnostic Accuracy for Liver Tumours Between the Combination of Contrast-enhanced Ultrasound and Contrast-enhanced Magnetic Resonance Imaging Versus Contrast-enhanced Computed Tomography and CEMRI
Brief Title: Comparing Diagnostic Accuracy for Liver Tumours Between the Combination of CEUS and CEMRI Versus CECT and CEMRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 201706079MIPA
Record Dates: First submitted 2017-08-27; First posted 2017-08-30 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2019-06

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sonazoid- CEUS+CEMRI or CECT+CEMRI (Experimental): Comparing Diagnostic Accuracy for Liver Tumours Between the Combination of CEUS and CEMRI Versus CECT and CEMRI
  Interventions: Diagnostic Test: Sonazoid- CEUS, CEMRI, CECT

INTERVENTIONS:
Diagnostic Test: Sonazoid- CEUS, CEMRI, CECT — Sonazoid- CEUS+CEMRI in a characterization of HCC, in comparison with CECT+CEMRI.

SUMMARY:
Hepatocellular carcinoma (HCC) is unique regarding diagnosis because the clinical diagnosis without pathology proof is accepted. The dynamic image, including contrast-enhanced computed tomography (CECT) and contrast-enhanced magnetic resonance image (CEMRI) were recognized in many guidelines for diagnosing the HCC. In contrast to the CT and MRI, ultrasound (US) with/without contrast is suggested by several societies as the sufficient surveillance modality. The contrast-enhanced ultrasound (CEUS) has aroused more attentions regarding the rapid improvement of contrast medium. In this study, the investigators conducted a prospective, single-center, open-label trial to compare the efficacy and safety of CEUS + CEMRI in characterizing HCC, in comparison with CECT + CEMRI.

DETAILED DESCRIPTION:
The liver cancers including hepatocellular carcinoma (HCC) resulted in more than 7,000 mortalities in Taiwan every year. HCC is unique regarding diagnosis because the clinical diagnosis without pathology proof is accepted. The dynamic image, including contrast-enhanced computed tomography (CECT) and contrast-enhanced magnetic resonance image (CEMRI) were recognized in many guidelines for diagnosing the HCC including Taiwan National Health insurance. Currently established guidelines endorse 3-phasic CT and MRI as first-line modalities. In contrast to the CT and MRI, ultrasound (US) with/without contrast is suggested by several societies as the most sufficient surveillance modality. However, the advantage of US in liver cirrhosis with regenerative nodules is only 32-65% in sensitivity.

The contrast-enhanced ultrasound (CEUS) has aroused more attentions regarding the rapidly improvement of contrast medium. In addition to Italian association for the study of the liver, the Japan society has documented CEUS as an integral part in the diagnosis algorism. Two phases, i.e. vascular phase and Kupffer phase, could be interpreted with second generation contrast agents, Sonazoid, for differentiating liver tumors. For liver tumor that failed to present washout phase in CECT or CEMRI, CEUS might be helpful because a tumor lack of contrast uptake in the Kupffer phase is favouring HCC. However, previous reports were confined to retrospective studies or small population, and more solid evidence is required to identify the diagnosis feasibility of CEUS with specific contrast agent.

In this study, the investigators conducted a prospective, single-center, open-label trial to compare the efficacy and safety of CEUS + CEMRI in characterizing HCC, in comparison with CECT + CEMRI. 60 patients with liver tumours no larger than 3cm in diameter will be enrolled, and tumour specimen will be obtained after imaging examination by tumour resection or biopsy. The primary endpoint is the sensitivity and specificity between the study groups, use the histology as reference diagnosis. The secondary endpoints include (1) the sensitivity and specificity of CEUS+CECT, CECT+CEMRI in differential diagnosis of liver tomours as malignant or benign, use the histology as reference diagnosis, (2) adverse effects, (3) vital signs (blood pressure, heart rate), and (4) laboratory values (the hematologic, renal and hepatic function change). Our exploratory endpoint is the detection rate of CEUS+CEMRI, CECT+CEMRI, use the histology as reference diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-70
2. All patients presented with newly diagnosed liver lesion(s) with initial impression of malignancy.
3. Lesions no larger than 3cm in diameter.
4. Signed and dated informed consent

Exclusion Criteria:

1. The lesion with previously documented histology
2. The lesion previously treated with Percutaneous Ethanol Injection, Radiofrequency Ablation, or Transarterial Chemoembolization
3. The lesion will not have histological confirmation after differential diagnosis
4. The subject had known hypersensitivity to any component of Sonazoid, including a history of allergies to eggs or egg products (i.e., manifested by full body rash, respiratory difficulty, oral or laryngeal swelling, hypotension or shock).
5. The subject was considered to be unsuitable to participate in the study by the investigator.
6. The subject was known to have a right-to-left shunt, severe pulmonary hypertension (pulmonary artery pressure >90 mmHg) or uncontrolled systemic hypertension.
7. The subject had a recent acute coronary syndrome or clinically unstable ischaemic cardiac disease, including: evolving or ongoing myocardial infarction, typical angina at rest within the last 7 days, significant worsening of cardiac symptoms within the last 7 days, recent coronary artery intervention or other factors suggesting clinical instability (e.g., recent deterioration of electrocardiogram, laboratory or clinical findings), acute cardiac failure, Class III/IV cardiac failure, or severe rhythm disorders.
8. The subject had adult respiratory distress syndrome, severe emphysema, pulmonary vasculitis, or a history of pulmonary emboli.
9. The subject had known thrombosis within the liver, or portal, or mesenteric veins.
10. The patient with iodine/Gd allergy, lower epidermal growth factor receptor level(<50), liver/renal dysfunction, and other condition that unsuitable to receive contrast
11. Pregnant and breastfeeding women

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2019-01-11 (Actual)

PRIMARY OUTCOMES:
The sensitivity and specificity of the blinded read of CEUS+CEMRI and CECT+CEMRI in characterization of HCC | up to 1 year
  the 95% two-sided confidence interval will be presented for both sensitivity and specificity in characterization of HCC

SECONDARY OUTCOMES:
The sensitivity and specificity of the blinded read of CEUS+CEMRI and CECT+CEMRI in differential diagnosis of liver tumours | up to 1 year
  the 95% two-sided confidence interval will be presented for both sensitivity and specificity in differential diagnosis of liver tumours

CONTACTS AND LOCATIONS:
Overall Officials: Kai-Wen Huang, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No